CLINICAL TRIAL: NCT03036891
Title: Naloxegol for Opioid-Related Gastroparesis: A Double-Blind Study With an Open Label Extension
Brief Title: Naloxegol for Opioid-Related Gastroparesis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24102
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Gastroparesis; Opioid Use
Keywords: Gastroparesis; Opioid-Induced; Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis | interventions — naloxegol; Tablets

STUDY DESIGN:
Intervention Model Description: The investigators have included a unique aspect of this study to better balance the benefits for patients participating in this randomized double-blind study in which half the patients receive a placebo agent. All patients in the treatment group and the placebo group will be invited to participate in the 4-week open-label extension for this study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Naloxegol 25 mg, oral tablet, daily for 4 weeks
  Interventions: Drug: Naloxegol 25 MG Oral Tablet [Movantik]
- Placebo Control (Placebo Comparator): Placebo Oral Tablet, 25 mg, oral tablet, daily for 4 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Naloxegol 25 MG Oral Tablet [Movantik] — Patients will be given the study drug (Movantik 25 mg).They will take this daily in the morning 1 hour before breakfast for four weeks.
  Other Names: Study
  Arms: Study Group
Drug: Placebo Oral Tablet — Patients will be given Placebo (Placebo 25 mg).They will take this daily in the morning 1 hour before breakfast for four weeks.
  Other Names: Control
  Arms: Placebo Control

SUMMARY:
The objective of this study is to evaluate the effects of naloxegol (a peripheral mu-opioid receptor antagonist [PAMORA]) in opioid-related gastroparesis on 1) symptoms of gastroparesis; 2) gastric emptying; and 3) pain control. The endpoints will be gastroparesis symptoms (PAGI-SYM), gastric emptying (GEBT), and pain control (McGill Pain Inventory). The hypothesis to be tested is that naloxegol improves symptoms of gastroparesis in patients who are taking opioids as well as improves their gastric emptying while maintaining control of patient's pain. This study will entail an initial double-blind, randomized, placebo-controlled, 4-week treatment period of naloxegol vs placebo in patients with opioid-related gastroparesis followed by a 4-week open label period to demonstrate the improvement in symptoms and gastric emptying with naloxegol.

DETAILED DESCRIPTION:
Medicines can delay gastric emptying and produce similar symptoms to gastroparesis. In particular, narcotic analgesics, can produce a gastroparesis picture, by delaying gastric emptying. The slowing effect of opioids on gastric, small bowel, and colonic motility has been well characterized. Unfortunately, many of these patients cannot stop their pain medications due to their underlying condition, such as back pain, fibromyalgia. On top of this, the narcotics can reduce the effectiveness of prokinetics agents used to treat gastroparesis, such as metoclopramide and domperidone. At this time, there is no good treatment for gastroparesis, especially for opioid-related gastroparesis.

Data suggests a relationship between opioid use and decreased gastric motility. Literature suggests that peripherally acting opioid agonist may provide relief in the instance of GI dysfunction (Holzer 2007). Movantik (Naloxegol) is an opioid agonist specifically designed to work outside of the central nervous system. Movantik (Naloxegol) can alleviate the adverse effects associated in chronic pain patients on opioid treatment - reduction of the undesired peripheral effects of opioids without disrupting analgesic effects. The use of Movantik (Naloxegol) has the potential to improve gastric dysmotility while preserving pain relief of the opioid analgesic.

The objective of this study is to evaluate the effects of naloxegol in opioid-related gastroparesis. This will be a randomized, double-blind study comparing Movantik 25 mg to placebo. The dose of Movantik is the dose that is currently FDA approved for opioid-induced constipation. The four-week study period is the duration of the phase 2b studies for Movantik for opioid-induced constipation in which the response rates were 60% and 35% with active treatment and placebo (Chey 2015).

The investigators have included a unique aspect of this study to better balance the benefits for patients participating in this randomized double-blind study in which half the patients receive a placebo agent. All patients in the treatment group and the placebo group will be invited to participate in the 4-week open-label extension for this study. This also serves to study the duration of the potential favorable effects of Movantik (Naloxegol) in this patient population as well as offering an extended time period to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-84, Males or Females
2. Daily use of narcotic analgesics for treatment of pain. Patients need to be on a stable daily dose of opiates for the last 4 weeks prior to enrollment
3. Patients with symptoms of gastroparesis with GCSI score (from the PAGI-SYM) of >2.0. These symptoms of gastroparesis must be present after starting opioid treatment.
4. Delayed gastric emptying based on previous scintigraphy (Percent gastric retention >60% at 2 hours and/or >10% retention at 4 hours
5. Signing informed consent prior to any study specific procedures

Exclusion Criteria:

1. Prior gastric resective surgery such as bariatric surgery, antrectomy.
2. Presence of severe renal impairment (CrCl<60 ml/min)
3. Presence of severe hepatic impairment - Child-Pugh Classification Class C, generally AST>200 or ALT>200 or Total bilirubin >3.0.
4. Other conditions besides gastroparesis that could potentially slow gastric emptying, such as untreated hypothyroidism.
5. Concomitants use of strong CYP 3A4 inhibitors (such as ketoconazole, diltiazem, erythromycin, clarithromycin), use of CYP3A4 inducer.
6. Use of NSAIDs and/or Plavix/Clopidogrel
7. Any prior use of Movantik (the study drug) or other opioid receptor antagonist (e.g., Relistor (methylnaltrexone), naltrexone, or naloxone) before the screening visit.
8. Patients with known cancer or cancer history within last 5 years prior to the screening visit.
9. Patients with GI obstruction and/or perforation or conditions with potential for GI perforation.
10. Patients with disruption to the blood-brain barrier;
11. Current use of a medication affecting gastric motility such as metoclopramide, domperidone, and erythromycin;
12. Pregnant women, females planning to become pregnant, and nursing mothers.
13. Women of childbearing potential who are unwilling to use contraceptives throughout the course of treatment
14. Subjects with severe co-morbidities (Cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, neurologic) based on PI's clinical judgment.
15. Active substance abuse.
16. History of major comorbid psychiatric conditions including mania and schizophrenia or severe current depression
17. At-risk populations, including prisoners and mentally challenged. Any condition or the patient is in a situation which may put him/her at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study (e.g., difficulty hearing, cognitive impairment)
18. Patients in which Movantik is clinically inadvisable
19. Subject unable to consent or is unwilling to provide informed consent

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Gastric Emptying (GE t-1/2) | 4 week
  Improvement in gastric emptying (GE t-1/2) compared to Placebo

SECONDARY OUTCOMES:
Daily Symptom Improvement using the GCSI-DD (Gastroparesis Cardinal Symptom Index-Daily Diary) | 4 weeks
  Improvements of gastroparesis symptoms using the GCSI-DD (Gastroparesis Cardinal Symptom Index-Daily Diary)
Symptom Improvement using PAGI-SYM | 4 weeks
  Improvements of gastroparesis symptoms using PAGI-SYM
Pain Management using the McGill Pain Inventory | 4 weeks
  Changes in pain control using the McGill Pain Inventory
Overall improvement in Gastric Emptying (GE t-1/2) | 8 week
  Improvement in gastric emptying (GE t-1/2) compared to Placebo
Quality of Life based on SF-36 | 4 weeks
  QOL score changes based on SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Henry Parkman, MD, Principal Investigator — Temple University Hospita
Locations (1):
- Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkman HP, Hasler WL, Fisher RS; American Gastroenterological Association. American Gastroenterological Association technical review on the diagnosis and treatment of gastroparesis. Gastroenterology. 2004 Nov;127(5):1592-622. doi: 10.1053/j.gastro.2004.09.055. PMID 15521026
- [Background] Abell TL, Bernstein RK, Cutts T, Farrugia G, Forster J, Hasler WL, McCallum RW, Olden KW, Parkman HP, Parrish CR, Pasricha PJ, Prather CM, Soffer EE, Twillman R, Vinik AI. Treatment of gastroparesis: a multidisciplinary clinical review. Neurogastroenterol Motil. 2006 Apr;18(4):263-83. doi: 10.1111/j.1365-2982.2006.00760.x. PMID 16553582
- [Background] Parkman HP, Yates K, Hasler WL, Nguyen L, Pasricha PJ, Snape WJ, Farrugia G, Koch KL, Calles J, Abell TL, McCallum RW, Lee L, Unalp-Arida A, Tonascia J, Hamilton F; National Institute of Diabetes and Digestive and Kidney Diseases Gastroparesis Clinical Research Consortium. Similarities and differences between diabetic and idiopathic gastroparesis. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1056-64; quiz e133-4. doi: 10.1016/j.cgh.2011.08.013. Epub 2011 Aug 24. PMID 21871247
- [Background] Anantharamu T, Sharma S, Gupta AK, Dahiya N, Singh Brashier DB, Sharma AK. Naloxegol: First oral peripherally acting mu opioid receptor antagonists for opioid-induced constipation. J Pharmacol Pharmacother. 2015 Jul-Sep;6(3):188-92. doi: 10.4103/0976-500X.162015. PMID 26312011
- [Background] Chey WD, Webster L, Sostek M, Lappalainen J, Barker PN, Tack J. Naloxegol for opioid-induced constipation in patients with noncancer pain. N Engl J Med. 2014 Jun 19;370(25):2387-96. doi: 10.1056/NEJMoa1310246. Epub 2014 Jun 4. PMID 24896818
- [Background] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003 Jul 1;18(1):141-50. doi: 10.1046/j.1365-2036.2003.01612.x. PMID 12848636
- [Background] Revicki DA, Rentz AM, Tack J, Stanghellini V, Talley NJ, Kahrilas P, De La Loge C, Trudeau E, Dubois D. Responsiveness and interpretation of a symptom severity index specific to upper gastrointestinal disorders. Clin Gastroenterol Hepatol. 2004 Sep;2(9):769-77. doi: 10.1016/s1542-3565(04)00348-9. PMID 15354277
- [Background] Revicki DA, Camilleri M, Kuo B, Norton NJ, Murray L, Palsgrove A, Parkman HP. Development and content validity of a gastroparesis cardinal symptom index daily diary. Aliment Pharmacol Ther. 2009 Sep 15;30(6):670-80. doi: 10.1111/j.1365-2036.2009.04078.x. Epub 2009 Jun 25. PMID 19558608
- [Background] Abell TL, Camilleri M, Donohoe K, Hasler WL, Lin HC, Maurer AH, McCallum RW, Nowak T, Nusynowitz ML, Parkman HP, Shreve P, Szarka LA, Snape WJ Jr, Ziessman HA; American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Consensus recommendations for gastric emptying scintigraphy: a joint report of the American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. J Nucl Med Technol. 2008 Mar;36(1):44-54. doi: 10.2967/jnmt.107.048116. Epub 2008 Feb 20. PMID 18287197
- [Background] Maranki JL, Lytes V, Meilahn JE, Harbison S, Friedenberg FK, Fisher RS, Parkman HP. Predictive factors for clinical improvement with Enterra gastric electric stimulation treatment for refractory gastroparesis. Dig Dis Sci. 2008 Aug;53(8):2072-8. doi: 10.1007/s10620-007-0124-7. Epub 2007 Dec 14. PMID 18080765
- [Background] Szarka LA, Camilleri M, Vella A, Burton D, Baxter K, Simonson J, Zinsmeister AR. A stable isotope breath test with a standard meal for abnormal gastric emptying of solids in the clinic and in research. Clin Gastroenterol Hepatol. 2008 Jun;6(6):635-643.e1. doi: 10.1016/j.cgh.2008.01.009. Epub 2008 Apr 14. PMID 18406670
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Culpepper-Morgan JA, Inturrisi CE, Portenoy RK, Foley K, Houde RW, Marsh F, Kreek MJ. Treatment of opioid-induced constipation with oral naloxone: a pilot study. Clin Pharmacol Ther. 1992 Jul;52(1):90-5. doi: 10.1038/clpt.1992.106. PMID 1623695
- [Background] Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003 Apr-Jun;35(2):253-9. doi: 10.1080/02791072.2003.10400007. PMID 12924748
- [Background] Peachey JE, Lei H. Assessment of opioid dependence with naloxone. Br J Addict. 1988 Feb;83(2):193-201. doi: 10.1111/j.1360-0443.1988.tb03981.x. No abstract available. PMID 3345396
- [Background] Tompkins DA, Bigelow GE, Harrison JA, Johnson RE, Fudala PJ, Strain EC. Concurrent validation of the Clinical Opiate Withdrawal Scale (COWS) and single-item indices against the Clinical Institute Narcotic Assessment (CINA) opioid withdrawal instrument. Drug Alcohol Depend. 2009 Nov 1;105(1-2):154-9. doi: 10.1016/j.drugalcdep.2009.07.001. Epub 2009 Aug 3. PMID 19647958
- [Background] Gandek B, Sinclair SJ, Kosinski M, Ware JE Jr. Psychometric evaluation of the SF-36 health survey in Medicare managed care. Health Care Financ Rev. 2004 Summer;25(4):5-25. PMID 15493441